CLINICAL TRIAL: NCT00002773
Title: A CLINICAL TRIAL FOR PANCREAS CANCER USING ACTIVE INTRALYMPHATIC IMMUNOTHERAPY WITH INTERFERON-TREATED PANCREAS CANCER TISSUE CULTURE CELLS, GMCSF, AND LOW-DOSE CYCLOPHOSPHAMIDE
Brief Title: Vaccine Therapy, Chemotherapy, and GM-CSF in Treating Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Vincent Medical Center - Los Angeles (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: SVMC-ONC-222P; CDR0000064749 (Registry Identifier: PDQ (Physician Data Query)); NCI-V96-0886
Record Dates: First submitted 1999-11-01; First posted 2004-04-29 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2007-04

CONDITIONS: Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Interferon-alpha; sargramostim; Cyclophosphamide

INTERVENTIONS:
Biological: allogeneic tumor cell vaccine
Biological: recombinant interferon alfa
Biological: sargramostim
Drug: cyclophosphamide

SUMMARY:
RATIONALE: Vaccines made from donated tumor cells treated with interferon alfa may make the body build an immune response to and kill pancreatic tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors may help a person's immune system recover from the side effects of chemotherapy. Combining these treatments may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining vaccine therapy using donated tumor cells treated with interferon alfa and radiation therapy and cyclophosphamide plus GM-CSF in treating patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility, toxicity, and antitumor effects of active specific intralymphatic immunotherapy with allogeneic pancreatic cancer cells treated with interferon alfa plus low-dose adjuvant systemic sargramostim (GM-CSF) and cyclophosphamide in patients with incurable pancreatic adenocarcinoma. II. Assess the immunologic and biologic correlates of this treatment regimen in these patients.

OUTLINE: Cultured allogeneic pancreatic cancer cells are incubated with interferon alfa for 72-96 hours. Autologous cell lines, if established, may be used as an alternative. The cells are irradiated immediately prior to use. Patients receive cyclophosphamide IV on day -3 and sargramostim (GM-CSF) subcutaneously on days 0-8. On day 0, patients receive viable tumor cells via dorsal pedal lymphatic cannulation. Treatment repeats every 2-4 weeks for a minimum of 8 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed every 2-4 months.

PROJECTED ACCRUAL: A total of 14 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the pancreas that is locoregionally active or metastatic and not amenable to cure or long-term control by surgery, radiotherapy, or chemotherapy No brain metastases refractory to irradiation or surgery

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-3 OR Karnofsky 60-100% Life expectancy: At least 3 months Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: No prior or concurrent significant cardiovascular disease Pulmonary: No prior or concurrent significant pulmonary disease Other: No AIDS HIV negative No prior or concurrent autoimmune disease No other concurrent major medical illness Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy Endocrine therapy: No concurrent chronic steroid therapy Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy Surgery: See Disease Characteristics Other: At least 4 weeks since other prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-05; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Wiseman, MD, FACP, Study Chair — St. Vincent Medical Center - Los Angeles
Locations (1):
- St. Vincent Medical Center - Los Angeles, Los Angeles, California, United States